CLINICAL TRIAL: NCT03230877
Title: The Evaluation of a Full Face Mask Seal for the Treatment of Obstructive Sleep Apnea
Status: Completed | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIA-223
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (2):
- Group A (Experimental): Participants will be randomized to receive either the "Improved Seal" or "Normal Seal" Toffee full face mask for a total of 7 ± 4 days from visit 1. At visit 2 they will return the first mask and be switched to the remaining mask for a total of 7 ± 4 days from visit 2.
  Interventions: Device: Toffee full face mask with 'Improved Seal'; Device: Toffee full face mask with 'Normal Seal'
- Group B (Experimental): Participants will be randomized to receive either the "Improved Seal" or "Normal Seal" Toffee full face mask for a total of 7 ± 4 days from visit 1. At visit 2 they will return the first mask and be switched to the remaining mask for a total of 7 ± 4 days from visit 2.
  Interventions: Device: Toffee full face mask with 'Improved Seal'; Device: Toffee full face mask with 'Normal Seal'

INTERVENTIONS:
Device: Toffee full face mask with 'Improved Seal' — Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1. Participants will be using the Improved Seal in this treatment arm.
Device: Toffee full face mask with 'Normal Seal' — Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1. Participants will be using the Normal Seal in this treatment arm.

SUMMARY:
The investigation is a prospective, randomized, single blinded, crossover study. The investigation is designed to evaluate the performance, comfort and ease of use of the F&P Trial Full Face Mask Seal amongst Obstructive Sleep Apnea (OSA) participants. A total number of 40-45 OSA participants will be recruited for the trial by the investigation site

DETAILED DESCRIPTION:
This study will involve three visits to the investigation site. During visit one participants will be randomized to, fitted with and issued with the first trial mask seal for use in- home for 7 ±4 days.

The participants will then come in to return the mask seal and be fitted and issued with the second trial seal for use in home for 7±4 days.

Visit Three will involve the participants returning the second trial seal and providing feedback.

ELIGIBILITY:
Inclusion Criteria:

* Adult (22+ years of age)
* Able to give informed consent
* Apnea hypopnea Index (AHI) ≥ 5 on diagnostic night
* Either prescribed Automatic positive airway pressure (APAP), Continuous positive airway pressure (CPAP) or Bi-level positive airway pressure (PAP) for OSA
* Fluent in spoken and written English
* Existing F&P full face mask user

Exclusion Criteria:

* Inability to give informed consent
* Participant intolerant to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or carbon Dioxide (CO2) retention
* Pregnant or may think they are pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials of Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
This investigation is to inform product development team. Results will inform product development on the future of the product.

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Seal Then Improved Seal: Participants will be randomized to the Normal Seal arm for a total of 7 ± 4 days from visit 1 and then will be crossed over to the Improved Seal arm for a total of 7 ± 4 days from visit 2.
- Improved Seal Then Normal Seal: Participants will be randomized to the Improved Seal arm for a total of 7 ± 4 days from visit 1 and then will be crossed over to the Normal Seal arm for a total of 7 ± 4 days from visit 2.
Period: Visit 1
Arm/Group | Normal Seal Then Improved Seal | Improved Seal Then Normal Seal
Started | 23 | 15
Completed | 23 | 15
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Normal Seal Then Improved Seal | Improved Seal Then Normal Seal
Started | 23 | 15
Completed | 23 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Population: Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1 and then crossed over to the other arm.
Arm/Group | Overall Population
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Trial Mask Seal Comfort
Description: Overall seal comfort determined from questionnaires- Subjective
Time Frame: 7 ± 4 days in-home
Measure: Count of Participants; unit: Participants
Groups:
- Toffee Full Face Mask With 'Improved Seal': Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1 and then crossed over to the other arm. Participants will be using a full face mask with the 'Improved Seal' in this treatment arm.
  Toffee full face mask with 'Improved Seal': Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1. Participants will be using the Improved Seal in this treatment arm.
- Toffee Full Face Mask With 'Normal Seal': Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1 and then crossed over to the other arm. Participants will be using a full face mask with the 'Normal Seal' in this treatment arm.
  Toffee full face mask with 'Normal Seal': Participants will be randomized to this arm for a total of 7 ± 4 days from visit 1. Participants will be using the Normal Seal in this treatment arm.
Arm/Group | Toffee Full Face Mask With 'Improved Seal' | Toffee Full Face Mask With 'Normal Seal'
Number analyzed (Participants) | 38 | 38
Participants
  Very comfortable | 16 | 13
  Comfortable | 16 | 19
  Neither comfortable nor uncomfortable | 2 | 1
  Uncomfortable | 3 | 3
  Very uncomfortable | 0 | 1
  N/A | 1 | 1

2. Primary Outcome: Trial Mask Seal Acceptability
Description: Preference for trial mask determined from questionnaires at the end of the trial - Subjective
Time Frame: 14 ± 4 days in-home
Measure: Count of Participants; unit: Participants
Groups:
- Total Trial Population: Participants will be randomized to one arm for a total of 7 ± 4 days from visit 1 and then crossed over to the other arm. After both seals are trialed, participant seal preference was collected
Arm/Group | Total Trial Population
Number analyzed (Participants) | 38
Participants
  Preferred "Improved seal" | 19
  Preferred "Normal seal" | 15
  No preference | 3
  N/A | 1

3. Secondary Outcome: Trial Mask Seal Treatment Performance - Objective
Description: Objective Apnea Hypopnea Index (AHI) data recorded from Positive airway pressure (PAP) device, compared to baseline AHI data
Time Frame: 7 ± 4 days in-home
Measure: Count of Participants; unit: Participants
Groups:
- Toffee Full Face Mask With "Improved Seal"; Toffee Full Face Mask With "Normal Seal": Participants will be randomized to one arm for a total of 7 ± 4 days from visit 1 and then crossed over to the other arm.
Arm/Group | Toffee Full Face Mask With "Improved Seal" | Toffee Full Face Mask With "Normal Seal"
Number analyzed (Participants) | 38 | 38
Participants
  Increased AHI | 10 | 6
  No change in AHI | 3 | 4
  Decreased AHI | 7 | 11
  N/A | 18 | 17

4. Secondary Outcome: Trial Mask Seal Usability
Description: Usability interview during first visit- Subjective
Time Frame: 1 hour day-time appointment
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask With 'Improved Seal' | Toffee Full Face Mask With 'Normal Seal'
Number analyzed (Participants) | 38 | 38
Participants
  Very easy | 28 | 26
  Easy | 8 | 7
  Neither easy nor difficult | 0 | 2
  Difficult | 0 | 1
  Very difficult | 0 | 0
  N/A | 2 | 2

5. Secondary Outcome: Trial Mask Seal Treatment Performance- Subjective
Description: Seal performance determined from questionnaires - Subjective
Time Frame: 7 ± 4 days in-home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask With 'Improved Seal' | Toffee Full Face Mask With 'Normal Seal'
Number analyzed (Participants) | 38 | 38
Participants
  Very good | 19 | 17
  Good | 11 | 12
  Neither good nor poor | 3 | 4
  Poor | 3 | 2
  Very poor | 1 | 2
  N/A | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all participants during the 2 month study period.
Arm/Group | Toffee Full Face Mask With 'Improved Seal' | Toffee Full Face Mask With 'Normal Seal'
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT03230877/Prot_SAP_000.pdf